CLINICAL TRIAL: NCT03761069
Title: Phase 1B Study of PTC299 in Relapsed/Refractory Acute Leukemias
Brief Title: Study of PTC299 (Emvododstat) in Relapsed/Refractory Acute Leukemias
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Sponsor terminated the study.
Sponsor: PTC Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PTC299-HEM-001-LEU
Record Dates: First submitted 2018-11-29; First posted 2018-12-03 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-01

CONDITIONS: Leukemia, Myeloid, Acute; AML
Keywords: Leukemia, Myeloid; Neoplasms by Histologic Type; Neoplasms; Dihydroorotate dehydrogenase (DHODH) inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Leukemia, Myeloid; Neoplasms by Histologic Type; Neoplasms | interventions — emvododstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- PTC299 (Experimental): PTC299 will be administered orally once daily (QD) for each 28-day cycle.
  Interventions: Drug: PTC299

INTERVENTIONS:
Drug: PTC299 — PTC299 will be administered per the treatment arm description
  Other Names: Emvododstat

SUMMARY:
This is an open-label, non-randomized, Phase 1b study to evaluate the safety, pharmacokinetics (PK) profiles, and preliminary evidence of antitumor activity of PTC299 and the metabolite, O-desmethyl PTC299, in participants with relapsed/refractory acute myeloid leukemia (AML) who have exhausted standard available therapies known to provide clinical benefit. The study is designed as a series of cohort-based dose escalations. For each cohort, a minimum of 3 evaluable participants with PK and safety data will be assessed. Additional participants will be recruited if additional PK data are needed to assess mean exposure based on the observed variability.

ELIGIBILITY:
Inclusion Criteria:

* Participant must have relapsed/refractory AML and exhausted standard available therapies known to provide clinical benefit.
* Subjects must be greater than or equal to 18 years of age.
* Subjects must have Eastern Cooperative Oncology Group (ECOG) performance status less than or equal to (≤) 2
* Women of childbearing potential must be willing to practice a highly-effective method of birth control for up to 50 days after the last dose of study drug.
* A man who is sexually active with a woman of childbearing potential and has not had a vasectomy must agree to use a barrier method of birth control during the study and for up to 50 days after the last dose of study drug.
* Subjects must be willing to participate to the study, have the ability to understand and adhere to study visit schedule and other protocol procedures, and be able and willing to sign a written informed consent form.

Exclusion Criteria:

Medical history:

* Women who are or plan to become pregnant, or who are currently breastfeeding.
* Persistence of any clinically relevant (Common Terminology Criteria for Adverse Events [CTCAE] Grade 2 or above) toxicities from previous therapy.
* Active alcohol or drug abuse.
* Previous drug-induced liver injury.

Cardiac assessments:

* Uncontrolled congestive heart failure, unstable angina pectoris.
* History or current evidence of a myocardial infarction during the last 6 months.
* QTc prolongation greater than (>) 500 milliseconds (msec) (Fridericia formula).
* Congenitally long QT syndrome or has received any marketed or experimental compound in the last 4 weeks or 5 half-lives (whichever is shorter) prior to entering the study with possible or known effects of QT prolongation. (If equivalent medication is not available, QTc will be closely monitored.)

Laboratory assessments:

* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) greater than or equal to (≥) 1 * upper limit of normal (ULN).
* Serum bilirubin ≥ 1 * ULN (except those known to have Gilbert's syndrome).
* Creatinine clearance ≤45 milliliters per minute (mL/min) (estimated by Cockcroft-Gault or by 24-hour urine collection).
* Any laboratory abnormality, which in the opinion of the investigator, places the participant at an unacceptably high risk for toxicities.

Gastrointestinal (GI) assessments:

* Liver malignancy (including metastases) or chronic liver disease.
* History of Gastrointestinal surgery or procedures or conditions that might interfere with the absorption or swallowing of the study drug.

Immunologic:

* Known hypersensitivity to study drug or its excipients.

Miscellaneous:

* Any sign of active uncontrolled infections; any severe chronic disease potentially interfering with the protocol, including human immunodeficiency virus (HIV) infection, or active hepatitis B or C or those with a positive screen for hepatitis A Immunoglobulin M (IgM).
* Any other malignancies within the past 2 years other than basal cell skin cancer or carcinoma in situ of the cervix.
* Participant concomitantly receiving any other investigational agents.
* Systemic chemotherapy within 2 weeks or investigational therapy within 5 half-lives prior to first dose of study drug, unless there is evidence of rapidly progressive disease (in which case the shorter washout of 2 weeks will be followed). For monoclonal antibodies, the washout from prior therapy will be 4 weeks, unless there is evidence of rapidly progressive disease, in which case, the shorter washout period of 2 weeks will be followed. Persistent chronic clinically significant toxicities from prior chemotherapy must not be >Grade 1. Use of hydroxyurea (Hydrea) is permitted up to 24 hours prior to start of study drug for control of proliferative disease. Hydrea treatment may be reinstated during study for control of proliferative disease, as needed, at the discretion of investigator.
* Participants with AML that has advanced with central nervous system (CNS) involvement.
* Participant is pregnant or breastfeeding or expecting to conceive or father children within the projected duration of the study.
* Participants receiving CYP2B6 substrates such as bupropion and methadone.
* Participants receiving strong CYP3A4 inducers such as carbamazepine, enzalutamide, mitotane, phenytoin, rifampin, and St. John's wort (hypericin) or drugs that are exclusively substrates of CYP3A4.
* Participant is receiving moderate or strong CYP3A4 inhibitors. (Note: This exclusion criterion is not applicable to subjects participating in sub-study where only subjects who are currently on/require antifungals [prophylaxis/treatment] will be enrolled)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2018-10-29 (Actual); Primary Completion 2021-12-28 (Actual); Study Completion 2021-12-28 (Actual)

PRIMARY OUTCOMES:
Number of Participants Who Discontinued Study Drug Due to Adverse Event (AE) | From Screening to 50 days post treatment

SECONDARY OUTCOMES:
Time to Maximum Plasma Concentration (Tmax) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Maximum Plasma Concentration (Cmax) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Area Under the Concentration-Time Curve (AUC) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Half-life (t1/2) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Estimate t1/2 of of both PTC299 and O-desmethyl PTC299 During 14-Day Washout Period | Day 29 through Day 42
Apparent Clearance (CL/F) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Apparent Volume of Distribution (Vz/F) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Accumulation Ratio (R) of both PTC299 and O-desmethyl PTC299 when PTC299 is Given as Tablet with Food | Days 1, 15, 28, 57, 71 and 99
Percentage of Participants Achieving Response Rate/Overall Response Rate Utilizing International Working Group (IWG) Response Criteria for AML | Up to 6 Months

CONTACTS AND LOCATIONS:
Locations (17):
- United States (17):
  - Rocky Mountain Cancer Center, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Henry Ford Health System, Detroit, Michigan
  - Rutgers, Cancer Institute of NJ, New Brunswick, New Jersey
  - Columbia, New York, New York
  - University of Rochester MC, Rochester, New York
  - Duke Cancer Center, Durham, North Carolina
  - Gabrail Cancer Center, Canton, Ohio
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Rhode Island, Miriam Hospital, Providence, Rhode Island
  - SCRI Tennessee Oncology, Nashville, Tennessee
  - Texas Oncology, P.A., Austin, Texas
  - Texas Oncology, P.A., Fort Worth, Texas
  - MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology, P.A. - San Antonio Medical Center, San Antonio, Texas
  - Swedish Cancer Institute, Seattle, Washington